CLINICAL TRIAL: NCT07400536
Title: A Phase III, Multicenter, Open-label, Randomized Controlled Clinical Study on the Treatment of Locally Advanced Cervical Cancer With Cadonilimab Combined With Chemotherapy Followed by Concurrent Chemoradiotherapy
Brief Title: A Clinical Study on the Treatment of LACC With Cadonilimab Combined With Chemotherapy Followed by CCRT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Akesobio (Industry)
Responsible Party: Principal Investigator, Guiling Li, PHD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-CC-001
Record Dates: First submitted 2026-02-02; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Cervical Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard concurrent chemoradiotherapy（CCRT） (Active Comparator): Accept standard concurrent chemoradiotherapy
  Interventions: Radiation: standard EBRT+Brachytherapy; Drug: Concurrent chemotherapy
- Cadonilimab+Induction chemotherapy+reduced-dose CCRT+Cadonilimab (Experimental): Undergo immune induction chemotherapy combined with reduced-dose radiotherapy and reduced-dose concurrent chemotherapy, and receive immune maintenance therapy after the completion of radiotherapy and chemotherapy.
  Interventions: Drug: Immune induction therapy; Radiation: Reduced dose radiotherapy; Drug: Dose reduction concurrent chemotherapy; Drug: Immunomaintenance therapy
- Cadonilimab+Induction chemotherapy+reduced-dose radiotherapy+Cadonilimab (Experimental): Undergo immune induction chemotherapy combined with reduced-dose radiotherapy, and receive immune maintenance therapy after the completion of radiotherapy and chemotherapy.
  Interventions: Drug: Immune induction therapy; Radiation: Reduced dose radiotherapy; Drug: Immunomaintenance therapy

INTERVENTIONS:
Radiation: standard EBRT+Brachytherapy — EBRT: 45-50.4Gy, Brachytherapy: 7Gy×4 or 6Gy
  ×5
  Arms: Standard concurrent chemoradiotherapy（CCRT）
Drug: Concurrent chemotherapy — Cisplatin 40mg/m2, qw×5
  Arms: Standard concurrent chemoradiotherapy（CCRT）
Drug: Immune induction therapy — Cadonilimab 10mg/kg q3w×2 + albumin paclitaxel 90mg/m2, qw×6+ cisplatin 25mg/m2, qw×6
  Arms: Cadonilimab+Induction chemotherapy+reduced-dose CCRT+Cadonilimab; Cadonilimab+Induction chemotherapy+reduced-dose radiotherapy+Cadonilimab
Radiation: Reduced dose radiotherapy — EBRT: 45-50.4Gy; Brachytherapy: 6Gy×4
  Arms: Cadonilimab+Induction chemotherapy+reduced-dose CCRT+Cadonilimab; Cadonilimab+Induction chemotherapy+reduced-dose radiotherapy+Cadonilimab
Drug: Dose reduction concurrent chemotherapy — cisplatin 25mg/m2, qw×5
  Arms: Cadonilimab+Induction chemotherapy+reduced-dose CCRT+Cadonilimab
Drug: Immunomaintenance therapy — Cadonilimab 10mg/kg q3w×9 or half a year
  Arms: Cadonilimab+Induction chemotherapy+reduced-dose CCRT+Cadonilimab; Cadonilimab+Induction chemotherapy+reduced-dose radiotherapy+Cadonilimab

SUMMARY:
This study mainly evaluated the efficacy and safety of Cadonilimab combined with chemotherapy followed by concurrent chemoradiotherapy versus standard concurrent chemoradiotherapy in the treatment of locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled, subjects had to meet all of the following criteria:

1. Female, aged 18-70 years (inclusive of cutoff values);
2. Histologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix;
3. Patients with stage IIB-IVA cervical cancer (FIGO stage 2018) who had not received any previous antineoplastic therapy;
4. At least one measurable lesion according to RECIST v1.1;
5. Eastern Cooperative Oncology Group (ECOG) performance-status score 0-1;
6. Have adequate organ function.

Exclusion Criteria:

Subjects were excluded from the study if they met any of the following criteria:

1. Distant metastatic disease (including inguinal lymph node metastasis and lymph node metastasis above the level of the superior edge of the L1 pyramid in the proximal cephalic region, according to FIGO 2018 stage IVB);
2. He had undergone total hysterectomy (removal of the corpus uteri and cervix);
3. Inability to undergo brachytherapy or refusal to undergo brachytherapy for reasons such as anatomical abnormalities;
4. Had received any previous antineoplastic therapy, including but not limited to surgery (except biopsy), radiotherapy, or systemic therapy (chemotherapy, immunotherapy, targeted therapy);
5. Had any condition that was deemed by other investigators to be ineligible for participation in the trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2028-07-18 (Estimated); Study Completion 2032-07-20 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) per RECIST 1.1 assessed by investigator(INV) | Up to approximately 55 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 | Up to approximately 55 months
  Assessed by investigators
Overall Survival (OS) | Up to approximately 55 months
  OS is defined as the time from randomization to death due to any cause.
Duration of Response (DOR) per RECIST 1.1 | Up to approximately 3 years
  Assessed by investigators
Time to Response (TTR) per RECIST 1.1 | Up to approximately 3 years
  Assessed by investigators
Disease Control Rate (DCR) per RECIST 1.1 | Up to approximately 3 years
  Assessed by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Guiling Li, PHD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: Undecided